CLINICAL TRIAL: NCT05306886
Title: Investigation of the Effect of Specially Designed and 3D Printed Insoles on Physical Activity Levels, Balance and Functional Performances
Brief Title: Investigation of the Effect of Specially Designed Insoles for Flat-footed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-BENLI-003
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Flat Foot [Pes Planus] (Acquired), Unspecified Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): ICB Special Insoles
  Interventions: Other: ICB Medical Insoles
- Control group (Active Comparator): ICB Insoles
  Interventions: Other: ICM Insoles

INTERVENTIONS:
Other: ICB Medical Insoles — After the foot analysis of the participants in the intervention group, special insoles will be designed in a computer program. In these insoles, 3-6 mm medial wedge support, 1-3 mm heel wedge support, 2-4 mm medial longitudinal arch support will be provided. These values will be determined according to the needs of each participant. A single physiotherapist will design all insoles. All drawings will be made by a single physiotherapist. After the design of the insoles is completed, insoles will be produced by transferring them to a Computer Numerical Control (CNC) machine. Ethyl vinyl acetate (EVA), the use of which has been found useful before, will be used as the material in the insoles molds. After processing, 1mm thick fabric will be used for the top coating. All insoles will be produced by the same physiotherapist.
  Arms: Intervention group
Other: ICM Insoles — As in the intervention group, insoles will be designed for the participants in the control group, processed by CNC machine and the production will be completed. Only 2mm medial longitudinal arch support will be given to the insoles of the people in this group.
  Arms: Control group

SUMMARY:
In our study, it was aimed to investigate the effect of insoles specially designed for each patient and printed with 3D printers on the physical activity levels, balance and functional performances of those patients.

DETAILED DESCRIPTION:
Our study, B.A.İ.B.Ü. İzzet Baysal Physical Therapy Training and Research Hospital and Fizyotermal Corp. It will be carried out as a dual center on individuals between the ages of 18-45 who apply to our clinic. It will be carried out by selecting 48 people who are suitable for the study among the flat-footed patients who applied to the clinics.

Patients will be evaluated before they start using the insoles, and immediately after using it , also after wearing the insoles for 8 weeks.

Patients will be randomized according to the order of their arrival at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* 1. Having a minimum 5 degree subtalar pronation angle while standing,
* 2. A minimum score of +6 from the Foot Posture Index (API) scale
* 3. Being between the ages of 18-45
* 4. Not having received any treatment from the foot area in the last 6 months
* 5. To have cognitive competence

Exclusion Criteria:

* 1. End of volunteering
* 2. Having a history of surgery of the lower extremity
* 3. Being an active athlete
* 4. Being pregnant or diagnosed with malignancy
* 5. Having a dysfunction such as severe neurological involvement, immobility, cooperation deficits that will limit physical activity
* 6. Lower extremity inequality greater than 1 centimeter (cm)
* 7. Having a different orthopedic disease that may affect lower extremity biomechanics
* 8. Receiving a different treatment for pes planus

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
The Physical Activity Assessment Questionnaire (IPAQ) Short Form | Eight weeks
  This form will be used to measure physical activity levels. comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity. Higher scores indicates better physical activity level.
Flamingo Balance Test and Y Balance Test | Eight weeks
  This will be applied for balance evaluation.To assess the ability to balance successfully on a single leg. A stopwatch, metal beam 50cm long, 5cm high and 3cm wide needed for test procedure. The total number of falls or loss of balance in 60 seconds is recorded. Scoring tables are available in the Eurofit Manual.

SECONDARY OUTCOMES:
Standing Long Jump Test | Eight weeks
  For functional performance Standing Long Jump test will be applied.The athlete stands behind a line marked on the ground with feet slightly apart. A two foot take¬off and landing is used, with swinging of the arms and bending of the knees to provide forward drive. The subject attempts to jump as far as possible, landing on both feet without falling backwards. Three attempts are allowed. The measurement is taken from take¬off line to the nearest point of contact on the landing (back of the heels). Record the longest distance jumped, the best of three attempts. The table below gives a rating scale for the standing long jump test for adults, based on personal experiences.
10 Meter Walk Test | Eight weeks
  For functional performance10 Meter Walk test will be applied. Patient's will be asked to walk 10 meter. Time is measured while patients walk.
Shuttle Running Test | Eight weeks
  For functional performance Shuttle Running Test will be applied. his test requires the person to run back and forth between two parallel lines as fast as possible. Set up two lines of cones 30 feet apart or use line markings, and place two blocks of wood or a similar object behind one of the lines.Two or more trails may be performed, and the quickest time is recorded. Results are recorded to the nearest tenth of a second.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Merkez, Turkey (Türkiye)